CLINICAL TRIAL: NCT06285448
Title: Feasibility of Lecanemab Registry and Clinical Outcome Measures
Status: Enrolling by invitation | Type: Observational
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Other Study IDs: A24-028
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease
Keywords: lecanemab
MeSH Terms: conditions — Alzheimer Disease | interventions — lecanemab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Alzheimer's disease: Patients with Alzheimer's disease eligible to receive lecanemab infusions at HealthPartners clinics and their care partners.
  Interventions: Drug: Lecanemab

INTERVENTIONS:
Drug: Lecanemab — Bi-weekly infusions of lecanemab [exposure].

SUMMARY:
Available FDA approved treatments for Alzheimer's disease (AD) temporary alleviate symptoms but have no bearing on overall disease progression. However, recent FDA approval of lecanemab (July 2023), a disease modifying therapy based on a phase 3 clinical trial demonstrated efficacy (cognitive) in persons with AD. Delaying the disease progression may impact not only the person living with dementia (PLWD), but also their Care Partners. It may provide the ability to achieve "life goals" as a family or may increase/reduce stress and burden on the family due to the complexity of the treatment regimen. Recent secondary analysis of this Phase 3 trial suggests quality of life showed less decline in PLWD and less increase in burden in Care Partners. The investigators propose to create a registry/database for persons living with dementia who receive lecanemab infusions at HealthPartners and their Care Partners. The investigators plan to test the feasibility of collecting outcomes data for specific patient and family focused outcomes, and outcomes that are typically not included in clinic. The outcome of this study will help in the overall goal of studying the impact of lecanemab in real-world settings in a larger cohort of PLWD and Care Partners.

ELIGIBILITY:
Inclusion Criteria:

* PLWD who are eligible to receive Lecanemab infusion at our clinics.
* Care Partner who provides care for the PLWD who are eligible to receive Lecanemab infusion at our clinics.
* Age >=18 years for PLWD and their care partners
* Provides informed consent prior to participation.

Exclusion Criteria:

* Unable to read and speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PLWD who are eligible to receive Lecanemab at HealthPartners clinics as standard of care, referred by clinic staff and their care partners.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of enrollment | 2 years
  Absolute number of potential care dyads (care partners and people living with dementia) contacted for recruitment and the number of those who consent and enroll.
Feasibility of completing visits | 3 months
  Number of enrolled participants completing the baseline and visit at 3 months.
Qualitative experience at 3 months | 3 months
  Summary of qualitative experience with lecanemab infusions at 3 months through survey and interviews .
Qualitative experience at 12 months | 12 months
  Summary of qualitative experience with lecanemab infusions at 12 months through survey and interviews .

CONTACTS AND LOCATIONS:
Overall Officials: Bhavani Kashyap, MBBS, PhD, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Neuroscience Center, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No